CLINICAL TRIAL: NCT03587597
Title: Esthetic Zone Socket Shield Technique With Immediate Temporization vs. Conventional Immediate Implant Placement With Immediate Temporization Randomized Clinical Trial
Brief Title: Socket Shield vs Conventional Immediate Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abd El Rahman, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03021984
Record Dates: First submitted 2018-06-09; First posted 2018-07-16 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Preservation of the Labial Bone
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket shield technique (Experimental): socket shield technique with immediate temporization
  Interventions: Procedure: socket shield technique
- conventional immediate implant (Active Comparator): conventional implant placement with immediate temporization
  Interventions: Procedure: conventional immediate implant placement with immediate temporization

INTERVENTIONS:
Procedure: socket shield technique — socket shield technique with immediate temporization
  Arms: socket shield technique
Procedure: conventional immediate implant placement with immediate temporization — conventional immediate implant placement with immediate temporization
  Arms: conventional immediate implant

SUMMARY:
eighteen implants will be placed in patients with non-restorable maxillary teeth in the aesthetic area.the recruited patients will be divided into two groups .group 1 will undergo socket shield technique with immediate temporization ,while group 2 will undergo conventional immediate implant placement with immediate temporization. to compare bone loss and aesthetic outcomes in the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable maxillary anterior teeth in the esthetic zone indicated for implant placement.
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
implant stability | immediately after implant placement
  implant stability will be measured using osstell device

SECONDARY OUTCOMES:
Amount of bone loss | after 3 month from implant insertion.
  Will be measured using linear measurements from CBCT

OTHER OUTCOMES:
pink aesthetic score | immediately after implant placement and three month later
  The gingival response to a anterior esthetic evaluation is assessed by the Pink Esthetic Score (PES) from clinical photography according to six variables scored from 0→2:
  1. Mesial & distal papillae,
  2. Keratinized gingiva,
  3. Curvature of the gingival margin,
  4. Level of the gingival margin,
  5. Root convexity(torque),
  6. Scar formation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided